CLINICAL TRIAL: NCT03999762
Title: Sperm Sample Preparation Protocol for Intrauterine Insemination (IUI)
Brief Title: Automated Sperm Sample Preparation Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanonc Inc. (Industry)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0619prep
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Density gradient sample prep (Active Comparator): Standard density gradient sample preparation
  Interventions: Device: sample prep
- Automated sample prep (Experimental): Automated experimental sample preparation
  Interventions: Device: sample prep

INTERVENTIONS:
Device: sample prep — Effectiveness of a sample preparation protocol

SUMMARY:
This clinical trial would be directed at determining the effectiveness of an innovative sperm sample preparation protocol for intrauterine insemination (IUI). The goal of the protocol would be to enable clinics not performing IUI to be able to perform IUI without requiring specialized training in sperm sample preparation.

DETAILED DESCRIPTION:
Nanonc proposes an automated system for sperm sample preparation that will take in raw ejaculate and output a purified sperm population in an IUI syringe in less than 15 minutes. The IUI syringe will be detachable from the rest of the system. During the 15 minutes, the clinician will not need to perform any actions; as the system will run all of the sample processing steps in an automated fashion. Furthermore, the system will have a footprint of a small desktop printer that is portable to be conveniently placed on a bench in clinical setting. A portable system that performs automated isolation of sperm from ejaculate will revolutionize sperm processing and increase access to sperm sample preparation. Additionally, the system will decrease cost, time and skill required to process sperm, and potentially improve outcomes for patients with low sperm counts. By increasing the yield and precision of sperm isolation and concentration techniques, the investigator's approach has the potential to offer this exact benefit by specifically providing the opportunity for some patients to try less invasive and less expensive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Any couple with doctor's order for IUI with density gradient centrifugation

Exclusion Criteria:

* Azoospermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-05-29 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Total motile sperm count | At the time of sperm preparation
  Total number of progressively motile sperm following sperm preparation
Percentage of patients with positive chemical pregnancy in each study group following IUI | 2 weeks after IUI
  Detection of hCG
Percentage of patients with positive clinical pregnancy in each study group following IUI | 6 to 7 weeks after IUI
  Detection of the fetal heartbeat by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Raheel Samuel, PhD, Principal Investigator — Nanonc Inc.

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.